CLINICAL TRIAL: NCT06653270
Title: Virtual Reality Simulation Training for Childbirth- a Cluster Randomised Crossover Study
Brief Title: Virtual Reality Birth Simulator
Acronym: ViVaDeX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: NUS-IRB-2020-606
Record Dates: First submitted 2024-09-09; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Medical Education; Normal Vaginal Delivery; Simulation Training; Virtual Reality
Keywords: Obstetrics; Labour; Vaginal delivery; Simulation training; Medical education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mannequin-based simulator (Active Comparator): Legacy PROMPT Flex® mannequin
  Interventions: Other: Mannequin-based simulator
- Virtual-reality simulator (Active Comparator): A in-house developed immersive virtual simulation of a normal vaginal delivery developed using a Unity Engine and installed in Oculus® Quest 2 head-mounted device
  Interventions: Other: Virtual reality simulator

INTERVENTIONS:
Other: Virtual reality simulator — A in-house developed immersive virtual simulation of a normal vaginal delivery developed using a Unity Engine and installed in Oculus® Quest 2 head-mounted device
  Other Names: ViVaDex
  Arms: Virtual-reality simulator
Other: Mannequin-based simulator — Legacy PROMPT Flex® mannequin
  Arms: Mannequin-based simulator

SUMMARY:
The investigators compared an in-house developed virtual reality simulator for normal vaginal deliveries with a legacy mannequin-based simulation in a cluster randomised study involving Year 4 medical students undergoing their Ob/Gyn clerkship with aims to compare pre- and post-simulation knowledge questionnaire score. As part of a cross-over component, the investigators will also compare feedback scores for each modality and the preferred modality. Ethical approval and waiver of consent has been obtained from the National University of Singapore Institutional Review Board, Reference Number 2020-606.

DETAILED DESCRIPTION:
Simulations training is an important aspect of procedural skills training. This is especially so for normal vaginal deliveries given its intimate and time sensitive nature. Medical students have to also compete with limited learning opportunities against other healthcare trainees in the labour ward. Thus, the need for simulation training has been extensively used in this area. Nevertheless, mannequin-based simulations are also limited in availability due to the need for expensive mannequins, skilled trainers, and suitable venues. The investigators developed a virtual reality normal vaginal delivery simulation (ViVaDex) based on the Oculus® Quest 2 retail Head Mounted Display and aim to compare this against legacy mannequin-based methods (PROMPT Flex®) via a a cluster randomised study involving Year 4 medical students undergoing their Obstetrics and Gynecology clerkship. The investigators would compare percentage correct scores pre- and post-simulation through an 11-item knowledge questionnaires and also conduct a six-domain feedback questionnaire. Due to a planned cross-over component, participants will be able to also state their preferred simulation modality.

Ethical approval and waiver of consent has been obtained from the National University of Singapore Institutional Review Board, Reference Number 2020-606.

Our statistical plan is to use two sample t-test to compare the improvement in pre- and post-simulation percentage correct scores between each modality and chi square testing to assess differences in the proportion who got each question correct. The feedback questionnaire scores will be compared between the VR and mannequin modalities using linear mixed modelling with teaching modality, period, and group being designated as main effects and presented as mean total feasibility scores with differences presented as adjusted mean difference with 95th centile confidence intervals (95% CI). Carryover effect will also be calculated as this is a cross-over study.

ELIGIBILITY:
Inclusion Criteria:

* Medical students undergoing their 4th year obstetrics and gynaecology clerkship

Exclusion Criteria:

* Declined to give consent or to have simulation videotaped

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Percentage improvement in knowledge scores | The time frame of involvement for each participant is 4 hours.
  Percentage of a knowledge quiz answered correctly before and after exposure to the first simulation device

SECONDARY OUTCOMES:
Mean scores from the feedback questionnaire | The time frame of involvement for each participant is 4 hours.
  Participants answered a Ffeedback Questionnaire after each simulation. A score was calculated based on this feedback. This feedback questionnaire 6 domain questionnaire comprising a mix of 14 positively- and negatively-framed questions that were scaled on a 5-point Likert scale with 1 indicating "strongly disagree" and 5 indicating "strongly agree".

CONTACTS AND LOCATIONS:
Locations (1):
- Yong Loo Lin School of Medicine, National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Percentage correct from the knowledge questionanire, type of questionnaire and the constituents.
Supporting Information: Study Protocol
Time Frame: 8th July 2022 to 30th Jul 2025